CLINICAL TRIAL: NCT01519687
Title: Open-Label, Inpatient Study of Levotofisopam 50 mg TID Administered for 7 Days to Men and Postmenopausal Women With Hyperuricemia and Gout
Brief Title: Study of Levotofisopam 50 mg Three Times a Day (TID) Administered for 7 Days on Hyperuricemia and Gout
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pharmos (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRS-TOFS-G201
Record Dates: First submitted 2012-01-24; First posted 2012-01-27 (Estimated); Last update posted 2012-01-27 (Estimated); Status verified 2012-01

CONDITIONS: Hyperuricemia; Gout
Keywords: hyperuricemia; gout; levotofisopam
MeSH Terms: conditions — Hyperuricemia; Gout | interventions — tofisopam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levotofisopam (Experimental): All patients will receive a single dose of 50 mg on Day 1, 50 mg three times a day (TID) on Days 2 through 6, and a single dose of 50 mg on Day 7. Each dose of study drug will be administered by authorized site personnel throughout the 7-day inpatient treatment period.
  Interventions: Drug: levotofisopam

INTERVENTIONS:
Drug: levotofisopam — 50 mg on Day 1, 50 mg TID on Days 2 through 6, and a single dose of 50 mg on Day 7
  Other Names: S-tofisopam

SUMMARY:
The purpose of this study is to determine whether levotofisopam is safe and effective in the treatment of hyperuricemia and gout.

DETAILED DESCRIPTION:
The primary objectives of this study are (1) to evaluate the safety and tolerability of levotofisopam in patients with hyperuricemia and gout, and (2) to evaluate the effect of treatment with levotofisopam on serum urate levels in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary, signed informed consent.
* Male or postmenopausal or surgically sterile females, 18 to 65 years of age, inclusive. Female participants must have been amenorrheic for a minimum of 12 months and must have a negative pregnancy test result within 3 days before administration of levotofisopam. Surgically sterile females are defined as those who have had a hysterectomy, bilateral ovariectomy, or bilateral tubal ligation. Male subjects must agree to practice a medically acceptable form of contraception for the duration of the study and for 30 days after receiving the last dose of levotofisopam.
* Physician diagnosis of gout with at least one gout flare in the last 6 months, at least one chronically swollen joint due to gout, or presence of a tophus.
* Serum urate level ≥ 8.0 mg/dL and ≤ 12.0 mg/dL after having stopped all urate-lowering therapy for at least 10 days. Serum urate level must also be > 7.7 mg/dL and ≤ 12.0 mg/dL on Day -3 and on Day -2.
* Willing and able to discontinue urate-lowering therapy starting at the screening visit (14-21 days before receiving study drug) through to the follow-up visit (up to 10 days after discharge from the study unit), for a total time off urate-lowering therapy of up to approximately 5 weeks.
* In the opinion of the investigator, able to participate in all scheduled evaluations, likely to complete all required tests, and likely to be compliant.
* Medications permitted for the treatment of non-excluded medical conditions (other than gout) must be at stable doses for at least 14 days prior to baseline.
* Permitted concurrent general medical conditions must be stable and well controlled.
* Written and oral fluency in the English language.

Exclusion Criteria:

* Previous treatment with racemic tofisopam (RS-tofisopam), levotofisopam (S-tofisopam), or dextofisopam (R-tofisopam).
* Known or suspected hypersensitivity to any benzodiazepine.
* History of two or more clinically significant drug allergies.
* Clinically significant infection within 30 days prior to screening or between screen and admission.
* History or presence of clinically significant medical disease that might compromise the study or be detrimental to the patient, such as hepatitis (patient excluded if hepatitis A was present within 2 years before screening or if there is any history of hepatitis B or C), human immunodeficiency virus (HIV) infection, uncontrolled diabetes mellitus, cirrhosis, active biliary disease (bile ducts or gallbladder), or moderate or severe chronic kidney disease (estimated glomerular filtration rate < 60 mL/min/1.73 m2).
* Presence of a gout flare during screening or the procedure window.
* History or presence of nephrolithiasis.
* History or presence of malignancy other than localized basal cell cancer, squamous cell skin cancer, or cancer in situ that has been resected within 5 years.
* Clinically significant head trauma with loss of consciousness within 10 years prior to screen.
* Myocardial infarction, congestive heart failure, or known coronary artery disease within 5 years prior to screen.
* Any history of cerebrovascular accident.
* History of seizure disorder other than a single childhood febrile seizure.
* Alcohol or psychoactive substance abuse or dependence, as defined by DSM-IV, within 1 year prior to screen, or alcohol use exceeding 21 units per week (on average) in the 3 months preceding screen.
* Used any tobacco- or nicotine-containing product more days than not within 30 days prior to screening or between screen and admission.
* Regular consumption (e.g., more days than not) of excessive quantities of caffeine-containing beverages (e.g., more than eight cups of coffee or equivalent per day) within 30 days prior to screening or between screen and admission.
* History of suicide attempt, any suicidal behavior within 6 months prior to screening or between screen and baseline, or, in the opinion of the investigator, clinically significant risk of suicide or violent behavior.
* History or presence of a clinically significant psychiatric disorder or symptom (e.g., delusions, hallucinations) that is likely to compromise the study (e.g., confound study results) or be detrimental to the patient.
* History of difficulty donating blood, or history or presence of clinically significant bleeding or hemorrhagic tendencies.
* Donation of blood or plasma within 90 days prior to screening or between screening and admission.
* Uncontrolled hypertension (systolic blood pressure > 160 mmHg and/or diastolic > 95 mmHg) or heart rate either < 50 BPM or > 100 BPM at any evaluation prior to the first dose of test drug.
* Pregnancy, lactation, a positive pregnancy test result during the screening or admission evaluation.
* A clinically significant abnormality on the screening physical examination, 12-lead electrocardiogram (ECG), or laboratory evaluations.
* A corrected QT (QTcF) value > 450 msec (males) or > 470 msec (females) at screening, admission (Day -3), or baseline (Day -1).
* Aspartate aminotransferase or alanine aminotransferase levels > 2 times upper limit of normal (ULN), alkaline phosphatase > 1.5 times ULN, creatinine outside the limits of normal, triglycerides > 500 mg/dL, or thyroid-stimulating hormone (TSH) levels greater than 6.0 µIU/L at screening, admission (Day -3), or Day -2.
* A finding of opiates, amphetamines, cocaine, cannabis, or phencyclidine on the urine drug screen (UDS). Any other positive UDS result must be discussed by the investigator and medical monitor prior to potentially allowing participation of the subject in the study.
* A positive HIV, hepatitis B, or hepatitis C test.
* Inability to take or tolerate colchicine for gout flare prophylaxis (0.6 mg QD or BID).
* Required use of any of the following from the screening visit through the follow-up visit: aspirin or other nonsteroidal antiinflammatory drugs (other than paracetamol, as noted below), diuretics, medications with known urate-lowering effects (including, but not limited to, fenofibrate, losartan, or vitamin C > 500 mg/day), or urate-lowering therapy other than levotofisopam.
* Dietary requirements inconsistent with the study unit's standardized diet.
* Body mass index ≥ 35.
* Use of any investigational treatment within 30 days prior to screening or between screen and admission.
* Use of any psychopharmacologic drug or substance within 7 days of screening or between screen and admission.
* Use of potent CYP3A4 inhibitors or potent CYP3A4 inducers within 7 days prior to screening or between screen and admission.
* An estimated 24-hour uric acid excretion > 1,000 mg/day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Percentage reduction in serum urate | Days 1-7
  The primary efficacy variable is the percentage reduction in serum urate from baseline to Day 7 on treatment with levotofisopam.

SECONDARY OUTCOMES:
Absolute reduction in serum urate from baseline | Days 1-7
  Secondary efficacy variables include absolute reduction in serum urate from baseline to Day 7 on treatment with levotofisopam, proportion of subjects with serum urate < 6 mg/dL on Day 7, change in fractional excretion of urate from baseline to Day 6, and change in 24-hour urinary uric acid from baseline to Day 6.

CONTACTS AND LOCATIONS:
Overall Officials: John S. Sundy, MD, PhD, Principal Investigator — Duke Clinical Research Unit
Locations (1):
- Duke Clinical Research Unit (DCRU), Durham, North Carolina, United States